CLINICAL TRIAL: NCT06575725
Title: A Phase 2 Study of Botensilimab, Balstilimab and Regorafenib in Patients With Microsatellite Stable Colorectal Cancer
Brief Title: Botensilimab, Balstilimab and Regorafenib or Botensilimab and Balstilimab for the Treatment of Advanced or Metastatic Microsatellite Stable Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Abandoned 9/23/24
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24074; NCI-2024-06706 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24074 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Advanced Colon Adenocarcinoma; Advanced Colorectal Adenocarcinoma; Advanced Rectal Adenocarcinoma; Metastatic Colon Adenocarcinoma; Metastatic Colorectal Adenocarcinoma; Metastatic Rectal Adenocarcinoma; Stage III Colon Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IV Colon Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Rectal Cancer AJCC v8
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms | interventions — balstilimab; Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm BB (botensilimab, balstilimab) (Experimental): Patients receive botensilimab IV over 60 minutes on day 1 of each cycle and balstilimab IV over 30 minutes on days 1, 15, and 29 of each cycle. Cycles repeat every 42 days for up to 2 cycles of botensilimab and up to 2 years of balstilimab in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and blood sample collection throughout the trial. Patients also undergo tumor biopsy during screening and on study.
  Interventions: Biological: Balstilimab; Procedure: Biopsy; Procedure: Biospecimen Collection; Biological: Botensilimab; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging
- Arm BBR (botensilimab, balstilimab, regorafenib) (Experimental): Patients receive botensilimab IV over 60 minutes on day 1 of each cycle, balstilimab IV over 30 minutes on days 1, 15, and 29 of each cycle, and regorafenib PO QD on days 1-7, 15-21, and 29-35 of each cycle or on days 1-5, 15-19, and 29-33 of each cycle. Cycles repeat every 42 days for up to 2 cycles of botensilimab and up to 2 years of balstilimab and regorafenib in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and blood sample collection throughout the trial. Patients also undergo tumor biopsy during screening and on study.
  Interventions: Biological: Balstilimab; Procedure: Biopsy; Procedure: Biospecimen Collection; Biological: Botensilimab; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Regorafenib

INTERVENTIONS:
Biological: Balstilimab — Given IV
  Other Names: AGEN 2034; AGEN-2034; AGEN2034
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Botensilimab — Given IV
  Other Names: AGEN 1181; AGEN-1181; AGEN1181; Anti-CTLA-4 Monoclonal Antibody AGEN1181
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Regorafenib — Given PO
  Other Names: BAY 73-4506 Monohydrate; BAY-73-4506 Monohydrate; Regorafenib Monohydrate; Stivarga
  Arms: Arm BBR (botensilimab, balstilimab, regorafenib)

SUMMARY:
This phase II trial studies how well the combination of botensilimab, balstilimab and regorafenib works compared to botensilimab and balstilimab in treating patients with microsatellite stable colorectal cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as botensilimab and balstilimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Regorafenib is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal protein that signals tumor cells to multiply. This helps to slow or stop the spread of tumor cells. The combination of botensilimab, balstilimab and regorafenib or botensilimab and balstilimab may be a safe and effective treatment for advanced or metastatic microsatellite stable colorectal cancer.

DETAILED DESCRIPTION:
COPRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of botensilimab, balstilimab and regorafenib (BBR) in microsatellite stable (MSS) metastatic colorectal cancer (mCRC) patients without metastatic liver lesions in the safety run-in. (Safety lead-in) II. Compare the overall response rate in microsatellite stable (MSS) metastatic colorectal cancer (mCRC) patients without metastatic liver lesions receiving botensilimab, balstilimab and regorafenib (BBR) versus botensilimab and balstilimab (BB), by treatment arm. (Phase II)

SECONDARY OBJECTIVES:

I. Estimate the overall survival in MSS mCRC patients without metastatic liver lesions receiving BBR and BB, by treatment arm.

II. Estimate the progression free survival in MSS mCRC patients without metastatic liver lesions receiving BBR and BB, by treatment arm.

III. Estimate the duration of response (DOR) in MSS mCRC patients without metastatic liver lesions receiving BBR and BB that experience a response to therapy, by treatment arm.

IV. Describe the safety of giving to BBR and BB to patients with MSS mCRC without metastatic liver lesions, by treatment arm.

EXPLORATORY OBJECTIVE:

I. Through the performance of baseline and on treatment biopsies and serial blood work (cytokines and flow cytometry), explore potential biomarkers of response to BBR and BB therapy given to MSS mCRC patients without metastatic liver lesions, by treatment arm.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM BBR: Patients receive botensilimab intravenously (IV) over 60 minutes on day 1 of each cycle, balstilimab IV over 30 minutes on days 1, 15, and 29 of each cycle, and regorafenib orally (PO) once daily (QD) on days 1-7, 15-21, and 29-35 of each cycle or on days 1-5, 15-19, and 29-33 of each cycle. Cycles repeat every 42 days for up to 2 cycles of botensilimab and up to 2 years of balstilimab and regorafenib in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) and blood sample collection throughout the trial. Patients also undergo tumor biopsy during screening and on study.

ARM BB: Patients receive botensilimab IV over 60 minutes on day 1 of each cycle and balstilimab IV over 30 minutes on days 1, 15, and 29 of each cycle. Cycles repeat every 42 days for up to 2 cycles of botensilimab and up to 2 years of balstilimab in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and blood sample collection throughout the trial. Patients also undergo tumor biopsy during screening and on study.

After completion of study treatment, patients are followed up at 30 and 90 days and then every 2-3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant
* In the phase II randomized portion of the study only, until two biopsies are obtained on ten patients receiving BBR and ten patients receiving BB: Agreement to biopsy of the same tumor at baseline and at 4 weeks

  * Agreement to biopsy of the same tumor at baseline and at 4 weeks

    * This applies only to patients with easily accessible tumors, where the risk of a biopsy is deemed acceptable. If a biopsy is determined to be unsafe patients will be exempt from this requirement
* Agreement to allow the collection of blood for correlatives at baseline, 1 week, 2 weeks, 4 weeks, 8 weeks, and at the time progressive disease
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 1
* Histologically or cytologically confirmed advanced or metastatic progressive proficient mismatch repair (pMMR)/MSS adenocarcinoma of the colon or rectum
* No active brain metastases or leptomeningeal metastases, except for patients who underwent definitive surgery or radiation without progression following repeat imaging (at least 4 weeks after the intervention) and were systemic steroids have been discontinued at least 2 weeks prior study treatment
* Known extended RAS and BRAF status, as per local standard of practice. Tumor mutation burden (TMB) and PD-L1 status will be collected when available but are not mandated for enrollment
* Patients must have progressed following exposure to all of the following agents in the advanced/metastatic setting OR in the neoadjuvant/adjuvant setting if disease recurred within 6 months of last treatment. Patients who were intolerant to prior systemic chemotherapy regimens are eligible if there is documented evidence of clinically significant intolerance despite adequate supportive measures

  * Fluoropyrimidines (capecitabine or 5-FU)
  * Irinotecan
  * Oxaliplatin
  * Anti-EGFR therapy if RAS and BRAF wild type with left colon primary
* Patients must have evidence of progression on or after the last treatment received and within 6 months prior to study enrollment
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy, excluding endocrinopathies stable on medication, stable neuropathy that is grade 2 or less, and alopecia
* Patients may not have metastatic liver disease defined as: No history of liver metastatic disease OR history of resected or ablated liver metastases without evidence of disease recurrence in the liver for at least 4 months before enrollment
* Total bilirubin ≤ 1.5 X upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN
* Alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 40 mL/min (measured or calculated using the Cockroft-Gault formula)
* Hemoglobin ≥ 9 g/dl
* Absolute neutrophil count (ANC) ≥ 1,500/µl
* Platelets ≥ 75,000/mm^3
* Albumin ≥ 3.0 g/dl
* Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 120 days after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men) OR have not been free from menses for > 1 year and ≥ 50 years of age (women only) OR amenorrheic for ≥ 2 years without a hysterectomy and bilateral oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation (women only) OR status is post-hysterectomy, bilateral oophorectomy, or tubal ligation (women only)

Exclusion Criteria:

* Prior allogeneic organ transplantation
* Prior immunotherapy with PD-1 or PD-L1 or CTLA-4 targeting agents
* Prior regorafenib
* Surgical intervention within 4 weeks prior to study treatment, except for minor procedures such as port placement
* Patients with a condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalent) within 14 days or another immunosuppressive medication within 30 days of the first dose of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Chemotherapy, radiation therapy, biological therapy, immunotherapy within 14 days or five half-lives (whichever is shorter for non-radiation therapy) prior to day 1 of protocol therapy
* Strong CYP3A4 inducers or CYP3A4 inhibitors within 14 days prior to day 1 of protocol therapy
* Patients unwilling to refrain from drinking grapefruit juice and taking St. John's Wort while on study
* Herbal medications other than cannabidiol (CBD) unless reviewed by the principal investigator (PI) and deemed to unlikely interact with study drugs
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 12 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥ III), or serious uncontrolled cardiac arrhythmia requiring medication
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Patients must not have uncontrolled hypertension as defined by systolic blood pressure (SBP) > 150mmHg or diastolic blood pressure (DBP) > 90mmHg despite optimal medical management. Patients whose blood pressure can be controlled medically are allowed to be rescreened once blood pressure (BP) is under control
* Active autoimmune disease or history of autoimmune disease that required systemic treatment within 2 years before starting treatment, i.e., with use of disease-modifying agents or immunosuppressive drugs
* History of acute thrombotic venous events in the last 30 days before enrollment. If within 30 days, the patient should be on anticoagulants and without symptoms
* Obstructive bowel symptoms related to unresected primary or carcinomatosis
* Inability to swallow and absorb oral tablets (such as but not limited to inability to swallow pills, malabsorption issues, ongoing nausea or vomiting)
* Non-healing wounds
* Symptomatic active bleeding
* Any evidence of current interstitial lung disease (ILD) or pneumonitis or a prior history of ILD or non-infectious pneumonitis requiring high-dose glucocorticoids
* History or current evidence of any condition, co-morbidity, therapy, any active infections, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator
* Known previous severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 10 days for mild or asymptomatic infections or 20 days for severe/critical illness prior to cycle 1 day 1 (C1D1)
* Uncontrolled infection with human Immunodeficiency virus (HIV). Patients on stable highly active antiretroviral therapy (HAART) with undetectable viral load and normal CD4 counts for at least 6 months prior to study entry are eligible. Serological testing for HIV at screening is not required
* Known to be positive for hepatitis B virus (HBV) surface antigen, or any other positive test for HBV indicating acute or chronic infection. Patients who are receiving or who have received anti-HBV therapy and have undetectable HBV deoxyribonucleic acid (DNA) for at least 6 months prior to study entry are eligible. Serological testing for HBV at screening is not required
* Known active hepatitis C virus (HCV) as determined by positive serology and confirmed by polymerase chain reaction (PCR). Patients on or who have received antiretroviral therapy are eligible provided they are virus-free by PCR for at least 6 months prior to study entry. Serological testing for HCV at screening is not required
* Dependence on total parenteral nutrition or intravenous hydration
* Clinically significant uncontrolled illness
* Concurrent non-colorectal second malignancy (present during screening) requiring treatment or history of a non-colorectal second primary metastatic malignancy within 2 years prior to the first dose of study treatment. Patients with history of prior early-stage basal/squamous cell skin cancer, low-risk prostate cancer eligible for active surveillance or noninvasive or in situ cancers who have undergone definitive treatment at any time are also eligible. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial after PI approval
* Females only: Pregnant or breastfeeding
* Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-01-28 (Estimated); Study Completion 2027-01-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (Safety lead in) | During cycle 1 (42 days)
  Assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Treatment related adverse event rates (Safety lead in) | During cycle 1 (42 days)
  Assessed by NCI CTCAE version 5.0.
Response rate (Phase II) RECIST | Up to 5 years after completion of study treatment
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 (primary) in microsatellite stable metastatic colorectal cancer patients without metastatic liver lesions receiving botensilimab, balstilimab and regorafenib versus botensilimab and balstilimab, by treatment arm. Will be summarized by number, and percentage, along with Clopper-Pearson exact binomial confidence intervals.
Response rate (Phase II) Immune-Modified RECIST | Up to 5 years after completion of study treatment
  Assessed by Immune-Modified RECIST (secondary) in microsatellite stable metastatic colorectal cancer patients without metastatic liver lesions receiving botensilimab, balstilimab and regorafenib versus botensilimab and balstilimab, by treatment arm. Will be summarized by number, and percentage, along with Clopper-Pearson exact binomial confidence intervals.

SECONDARY OUTCOMES:
Overall survival | From enrollment to death as a result of any cause or being censored at their last contact, assessed up to 5 years after completion of study treatment
  Will be estimated by the Kaplan-Meier method and calculated with 95% confidence intervals (CIs).
  Will be summarized by number, and percentage, along with Clopper-Pearson exact binomial confidence intervals.
Progression free survival | From enrollment to disease progression/relapse or death as a result of any cause, whichever occurs first, assessed up to 5 years after completion of study treatment
  Will be estimated by the Kaplan-Meier method and will be calculated with 95% CIs.
  Will be summarized by number, and percentage, along with Clopper-Pearson exact binomial confidence intervals.
Duration of treatment response | Up to 5 years after completion of study treatment
  Defined as time to progression or death, starting at the time when a response is experienced.
Incidence of adverse events | Up to 90 days after completion of study treatment
  Defined as toxicity, graded according to the NCI CTCAE v5.0. Toxicity data will be summarized in frequency tables by category and grade to evaluate the safety profile of the combination therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Marwan G Fakih, Principal Investigator — City of Hope Medical Center